CLINICAL TRIAL: NCT03568552
Title: Patient Decision Aid for Medication-Assisted Treatment for Opioid Use Disorder
Brief Title: Patient Decision Aid for Opioid Use Disorder
Acronym: PtDA-MAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Yih-Ing Hser, Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OPIOD1.1
Record Dates: First submitted 2018-06-03; First posted 2018-06-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder (OUD); Medication Assisted Therapy (MAT); Patient Decision Aid; Medication Treatment for Opioid Use Disorder (MOUD)
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The Patient Decision Aid for Medication Assisted Therapy (PtDA-MAT) will be tested by patients and clinicians during actual visits with OUD patients to assess its acceptability and effectiveness. We will track patients receiving PtDAT-MAT using their clinical and administration data over a 24-month period to assess outcomes associated with PtDAT-MAT. Participating clinics will be randomly selected in sequence to implement the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Decision Aid (Experimental): Participating clinics (and their patients) will be randomly selected to implement the intervention, at which time their patients will receive Patient Decision Aid for Medication Assisted Treatment for opioid use disorder.
  Interventions: Behavioral: Patient Decision Aid
- Prior to intervention (No Intervention): All participating clinics will start with a baseline period without the intervention. The clinics and their patients will remain in the no intervention condition until randomly selected to crossover to receive the intervention.

INTERVENTIONS:
Behavioral: Patient Decision Aid — PtDA-MAT will provide information on MAT treatment options and pros and cons of each treatment option, and will assess patients' preferred options.
  Arms: Patient Decision Aid

SUMMARY:
The aim of the study is to test the effectiveness of the Patient Decision Aid for Opioid Use Disorder (PtDA-MAT) by conducting a stepped-wedge cluster-randomized trial in CA H&SS (stratified by rural vs. non-rural areas) for adults with OUD. Patient outcomes will be tracked by (1) personal assessments (baseline, 3 months, and 6 months): drug use, overdose, healthcare utilization, and (2) clinical and administrative records (over approximately 24 months): drug treatment status and retention, physical and mental health diagnoses, arrest, incarceration, controlled substance use, and mortality. Multilevel models will be applied to test the intervention effects, controlling for possible temporal trends.

DETAILED DESCRIPTION:
In response to RFA-DA-18-005 (Expanding Medication Assisted Treatment for Opioid Use Disorders in the Context of the SAMHSA Opioid STR Grants, R21/R33), this project will develop and test a patient decision support tool called Patient Decision Aid for Medication-Assisted Treatment (PtDA-MAT) for use in the CA H&SS. The PtDA-MAT is designed to (1) improve patient knowledge and involvement and to subsequently improve treatment adherence and outcomes and (2) to support clinicians in informing and communicating with their patients with OUD along a continuum of care. The 3 year project will assess the effectiveness of the PtDA-MAT in a stepped-wedge cluster-randomized trial in CA H&SS (stratified by rural vs. non-rural areas) for adults with OUD. Patient outcomes will be tracked by (1) personal assessments (baseline, 3 months, and 6 months): drug use, overdose, healthcare utilization, and (2) clinical and administrative records (over an average of 24 months): drug treatment status and retention, physical and mental health diagnoses, arrest, incarceration, controlled substance use, and mortality. Multilevel models will be applied to test the intervention effects, controlling for possible temporal trends.

ELIGIBILITY:
Inclusion Criteria:

* Opioid Use Disorder diagnosis and agreement to follow study procedures (including permission to share medical records and other administrative records)

Exclusion Criteria:

* Significant or unstable medical or psychiatric illness that may interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7554 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Treatment Retention | 24 months
  Treatment retention will be defined as time from initial treatment admission to either MAT discontinuation or most recent clinic visit followed by 2 months gap in treatment
Opioid Use at 3 months | 3 months
  Self-reported days of opioid use in past 4 weeks
Opioid Use at 6 months | 6 months
  Self-reported days of opioid use in past 4 weeks

SECONDARY OUTCOMES:
Substance Use | 24 months
  Opioid-negative urine drug screen results (as collected by clinics as part of routine care) and other substance use per self-report (e.g., cannabis, benzodiazepines, cocaine, amphetamines)
Treatment Adherence | 24 months
  Treatment Adherence defined as proportion of clinic visits attended
Mortality | 24 months
  National Death Index maintained by the national Centers for Disease Control and Prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Ing Hser, Ph.D., Principal Investigator — University of California, Los Angeles; Larissa Mooney, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Integrated Substance Abuse Programs, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided